CLINICAL TRIAL: NCT02350075
Title: Clinical Success of Short Dental Implants Alone and Standard Dental Implants Combined With Osteotome Sinus Floor Elevation in Posterior Maxillae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Medical Doctor, Department of oral and maxillofacial implants, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012CB933600
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Jaw, Edentulous, Partially
Keywords: short implants; sinus floor elevation; randomized controlled trial
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short implants group (Experimental): Patients receive short dental implants installation (6mm) without additional augmentation procedures.
  Interventions: Procedure: Dental implants installation
- Standard implants with OSFE group (Other): Patients receive standard dental implants installation (10mm) combined with osteotome sinus floor elevation.
  Interventions: Procedure: Dental implants installation; Device: Osteotome Sinus floor elevation

INTERVENTIONS:
Procedure: Dental implants installation — Dental implants installation is a procedure to insert dental implants into alveolar bone.
Device: Osteotome Sinus floor elevation — Osteotomes with different diameters are specially-designed device to vertically increase the bone volume in atrophic maxilla.
  Arms: Standard implants with OSFE group

SUMMARY:
The aim of this study is to determine the clinical success of short implants (6mm) alone and standard implants (10mm) combined with sinus floor elevation in atrophic maxilla.

DETAILED DESCRIPTION:
Implant treatment in posterior maxilla is commonly faced with great challenges due to the limited residual bone height and poor bone quality. Efforts have been made to allow successful implant treatment in atrophic posterior maxillae.Osteotome sinus floor elevation (OSFE) has been proven to be a predictable surgical procedure to vertically increase the bone volume in atrophic maxilla.On the other hand, short implants (intra-bony length of 8mm or less) are being increasingly used in extremely resorbed maxilla to avoid additional surgical trauma and expense.However, still limited randomized controlled trials have compared the clinical success of short implants and standard implants combined with OSFE.

This study is designed as a prospective randomized controlled clinical study. We plan to enroll 180 patients in need of dental implant treatment in posterior maxilla. All patients will sign the informed consent form before treatment. The study is approval by the Ethics Committee of Shanghai Ninth People Hospital, China. The clinical component of the study will be initiated in May 2015 at the Department of Oral and Maxillofacial Implantology, Shanghai Ninth People Hospital, Shanghai Jiao-Tong University, China.

A block randomization sequence will be used to assign eligible patients to three groups: Group 1: short implants (6mm) alone; Group 2: standard implants (10mm) combined with OSFE. The assignment will be concealed from the clinical operators until the beginning of implant surgery. The outcome examiners and patients will be kept blinded to the assignment.

The required sample size is calculated based on the primary outcome parameter, implant survival rate. A recent study (Rossi et al. 2016) compared survival rate of short implants and standard implants (Survival rate: 86.7% VS 96.7%). If α=0.05, and 1-β =0.8, a sample size of n=116 per group is required. Assuming a drop-out rate of 10%, 125 patients per group will be required. The total required sample size will thus be n=250.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria are applied:

* age≧18 years, partial edentulism in posterior maxilla for at least three months from tooth loss,
* residual bone height range from 6-8mm,
* sufficient bone width in edentulous region.

Exclusion Criteria:

The patients will be excluded on the basis of:

* heavy smoker (>10 cigarettes per days),
* uncontrolled diabetes mellitus or other systemic diseases,
* uncontrolled periodontal infection,
* insufficient bone quality to achieve implant stability and
* previous implant installation or bone grafting at surgical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-03-01; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Implants survival rate | 1 year after implant placement
  Survival rate is defined by percentage of dental implants that remained in situ with or without modifications.

SECONDARY OUTCOMES:
Marginal bone loss | 1 year after implant placement
  Alveolar bone loss around dental implants during the observation period
Complication rate | 1 year after implant placement
  Both biological and mechanical complications will be recorded
Patient-reported outcome (100-mm visual analogue scale (VAS) | 10 minutes after implant surgery
  Patients will be asked to give their answer regarding surgical comfort using a 100-mm visual analogue scale (VAS) with word "very dissatisfied" to "very satisfied" on the left and right end respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Jun-Yu Shi, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Mangano FG, Shibli JA, Sammons RL, Iaculli F, Piattelli A, Mangano C. Short (8-mm) locking-taper implants supporting single crowns in posterior region: a prospective clinical study with 1-to 10-years of follow-up. Clin Oral Implants Res. 2014 Aug;25(8):933-40. doi: 10.1111/clr.12181. Epub 2013 Apr 28. PMID 23621393
- [Background] Lai HC, Si MS, Zhuang LF, Shen H, Liu YL, Wismeijer D. Long-term outcomes of short dental implants supporting single crowns in posterior region: a clinical retrospective study of 5-10 years. Clin Oral Implants Res. 2013 Feb;24(2):230-7. doi: 10.1111/j.1600-0501.2012.02452.x. Epub 2012 Apr 2. PMID 22469075
- [Background] Tan WC, Lang NP, Zwahlen M, Pjetursson BE. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. Part II: transalveolar technique. J Clin Periodontol. 2008 Sep;35(8 Suppl):241-54. doi: 10.1111/j.1600-051X.2008.01273.x. PMID 18724853
- [Background] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Background] Thoma DS, Haas R, Tutak M, Garcia A, Schincaglia GP, Hammerle CH. Randomized controlled multicentre study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures. Part 1: demographics and patient-reported outcomes at 1 year of loading. J Clin Periodontol. 2015 Jan;42(1):72-80. doi: 10.1111/jcpe.12323. Epub 2014 Dec 26. PMID 25418606
- [Derived] Zhang XM, Shi JY, Gu YX, Qiao SC, Mo JJ, Lai HC. Clinical Investigation and Patient Satisfaction of Short Implants Versus Longer Implants with Osteotome Sinus Floor Elevation in Atrophic Posterior Maxillae: A Pilot Randomized Trial. Clin Implant Dent Relat Res. 2017 Feb;19(1):161-166. doi: 10.1111/cid.12435. Epub 2016 Jul 8. PMID 27389435
- [Derived] Shi JY, Gu YX, Qiao SC, Zhuang LF, Zhang XM, Lai HC. Clinical evaluation of short 6-mm implants alone, short 8-mm implants combined with osteotome sinus floor elevation and standard 10-mm implants combined with osteotome sinus floor elevation in posterior maxillae: study protocol for a randomized controlled trial. Trials. 2015 Jul 30;16:324. doi: 10.1186/s13063-015-0853-4. PMID 26223254